CLINICAL TRIAL: NCT05315102
Title: To Investigate the Effects of Three Weeks of Intensive Chiropractic Care When Added to Usual Care for Children With Cerebral Palsy.
Brief Title: Effects of Intensive Chiropractic Care to Usual Care for Children With Cerebral Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/01285 Imran Amjad
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Research
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A registered chiropractor will assess the entire spine, and both sacroiliac joints will be assessed for vertebral subluxation by a registered chiropractor. The clinical indicators that will be used to assess the function of the spine before spinal adjustment intervention include assessing for joint tenderness to palpation manually palpating for a restricted intersegmental range of motion, assessing for palpable asymmetric intervertebral muscle tension, and any abnormal or blocked joint play and end-feel of the joints.
  Interventions: Other: Chiropractic Care; Other: Physical therapy intervention
- Control group (Sham Comparator): The participants head and/or spine will be moved in ways that include passive and active movements, similar to what is done when assessing the spine by a chiropractor.No spinal adjustment will be performed during any control intervention.
  Interventions: Other: Sham intervention; Other: Physical therapy intervention

INTERVENTIONS:
Other: Sham intervention — The participants head and/or spine will be moved in ways that include passive and active movements, similar to what is done when assessing the spine by a chiropractor. The sham intervention will also include the participants moving into adjustment setup positions similar to how the chiropractor would typically set up a patient with no joint pre-loading or adjustive thrust
  Arms: Control group
Other: Chiropractic Care — A registered chiropractor will assess the entire spine, and both sacroiliac joints will be assessed for vertebral subluxation by a registered chiropractor. The clinical indicators that will be used to assess the function of the spine before spinal adjustment intervention include assessing for joint tenderness to palpation manually palpating for a restricted intersegmental range of motion, assessing for palpable asymmetric intervertebral muscle tension, and any abnormal or blocked joint play and end-feel of the joints.
  Arms: Experimental group
Other: Physical therapy intervention — The standardized treatment protocol will be provided according to the guidelines, which will include various modalities and treatment approaches, including stretching exercises; massage; strengthening exercises of weak muscles, weight-bearing, balance (static and dynamic) and gait training; electrical stimulation; treadmill use; and endurance training for the improvement of gait, motor function, strength and functional mobility in Cerebral Palsy children, where Conventional Therapy will be provided according to the respective needs of the individual patient.

SUMMARY:
To determine the effects of chiropractic care on spasticity, functional outcomes and quality of life in spastic cerebral Palsy children.

ELIGIBILITY:
Inclusion Criteria:

Participants will be recruited into the study according to the following criteria.

* Both gender (Male and Female).
* Age between 2 to 15 years.
* Spastic Cerebral Palsy children.

Exclusion Criteria:

Participants will be excluded from the study according to the following criteria.

* Cerebral Palsy children due to Traumatic Brain Injury.
* Patients having cognitive impairments.
* Patients having associated Neurological Pathologies.
* Patients who are unable to follow treatment plan.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure | 3 weeks
  The gross motor function measure is a standard instrument that measures the change in motor function with time in Cerebral palsy subjects. It assesses the number of motor tasks a child can perform.
  A scoring key of 0 - does not initiate, 1 - initiates, 2 - partially completes, and 3 - completed, is used. the higher score, the greater is Gross motor function.
Trunk Control Measurement Scale (TCMS) | 3 weeks
  TCMS is an extended version of the trunk impairment scale with a total score of 58, which assesses the quality of static and dynamic trunk control.
  The maximum value for the total TCMS is 58 points (20 for the category 'static sitting balance', 28 for 'selective movement control', and 10 for 'dynamic reaching'). A higher TCMS score indicates better performance in trunk control.
Melbourne Assessment of Unilateral Upper Limb Function (MUUL) | 3 weeks
  Melbourne Assessment of Unilateral Upper Limb Function (MUUL) is considered as one of the reliable tools to measure upper limb function. It consists of 16-items to measure the quality of unilateral upper limb function.
  Scoring is completed across the 30 score items using a three, four or five-point scale and individually defined scoring criteria. Item scores relating to each element of movement measured are summed within the corresponding sub-scale.
Canadian Occupation Performance Measure (COPM) | 3 weeks
  It is a client-centred outcome measure that helps the client to identify occupational performance issues and rates performance and satisfaction pre and post-intervention.
  Total scores are calculated by adding together the performance or satisfaction scores for all problems and dividing them by the number of problems. At reassessment, the client scores each problem again for performance and satisfaction.
Cerebral Palsy Quality Of Life scale (CP-QOL) | 3 weeks
  The CP-QOL-child is a condition-specific QOL questionnaire designed for children with CP. QOL is broadly defined as a subjective multidimensional concept for assessing a person's wellbeing across numerous life indicators.
  The greater the score, the better is the quality of life.
Smartphone app for gait and Balance Assessment | 3 weeks
  This embedded inertial sensor-based smartphone application can provide a valid and reliable estimation of several gaits and balance parameters. The smartphone app for gait and balance assessment will be used on the subject who can walk independently.

CONTACTS AND LOCATIONS:
Overall Officials: IMRAN AMJAD, PhD, Principal Investigator — Riphah International University
Locations (1):
- National Institute of rehabilitation medicine., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No